CLINICAL TRIAL: NCT01711489
Title: A Phase 1, Open-Label, Sequential Study of the Effect of Multiple Doses of Isavuconazole on the Pharmacokinetics of a Single Dose of Mycophenolate Mofetil in Healthy Adult Subjects
Brief Title: A Study to Assess the Effect of Multiple Doses of Isavuconazole on the Pharmacokinetics of a Single Dose of Mycophenolate Mofetil in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 9766-CL-0030
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Healthy Subjects; Pharmacokinetics of Isavuconazole; Pharmacokinetics of Plasma Mycophenolic Acid (MPA); Pharmacokinetics of Plasma Phenolic Glucuronide of MPA (MPAG)
Keywords: isavuconazole; mycophenolate mofetil (MMF); BAL8557; BAL4815; healthy volunteers; Mycophenolic acid (MPA); Phenolic glucuronide of MPA (MPAG); CellCept
MeSH Terms: interventions — isavuconazole; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- isavuconazole and mycophenolate mofetil (Experimental): Single dose of MMF on Day 1, isavuconazole three times daily (TID) on Days 9 and 10, isavuconazole once daily (QD) Days 11-16, a single dose of MMF on Day 13
  Interventions: Drug: isavuconazole; Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: isavuconazole — oral
  Other Names: BAL4815
Drug: Mycophenolate mofetil — oral
  Other Names: CellCept, MMF

SUMMARY:
The purpose of this study is to assess the effect of multiple doses of isavuconazole on the pharmacokinetics (PK) of mycophenolate mofetil (MMF) after single dose administration. Safety and tolerability of isavuconazole will be assessed alone and in combination with MMF.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body weight of at least 45 kg and has a body mass index (BMI) of 18 to 32 kg/m2, inclusive.
* Results for aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must be ≤ 1.5 mg/dL
* The female subject agrees to sexual abstinence, or is surgically sterile, postmenopausal (defined as at least 2 years at Screening without menses), or using a medically acceptable double barrier method (e.g. spermicide and diaphragm, or spermicide and condom) to prevent pregnancy and agrees to continue using this method from Screening until 5 weeks after the follow-up visit at the end of the study; and is not lactating or pregnant as documented by negative pregnancy tests at Screening and Day -1.
* The male subject agrees to sexual abstinence, is surgically sterile, or is using a medically acceptable method to prevent pregnancy and agrees to continue using this method from Screening until 5 weeks after the follow-up visit at the end of the study

Exclusion Criteria:

* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of Long QT syndrome (suggested by sudden death of a close relative at a young age due to possible or probable cardiac causes).
* The subject has a history of tuberculosis or exposure to anyone known or suspected to have tuberculosis or any illness that might confound the results of the study or pose additional risk in administering study drug to the subject.
* The subject has a positive result for hepatitis C antibodies, hepatitis B surface antigen, or QuantiFERON®-TB Gold test at Screening or is known to be positive for human immunodeficiency virus (HIV).
* The subject has a known or suspected allergy to any of the components of the trial products including mycophenolate mofetil (MMF) or the azole class of compounds, or a history of multiple and/or severe allergies to drugs or foods, or a history of severe anaphylactic reactions.
* The subject is a smoker (any use of tobacco or nicotine containing products) within 6 months prior to Screening.
* The subject has had treatment with prescription drugs or complementary and alternative medicines within 14 days prior to Day -1, or over-the-counter medications within 1 week prior to Day -1, with the exception of acetaminophen up to 2 g/day.
* The subject has a recent history (within the last 2 years) of drug or alcohol abuse, as defined by the investigator, or a positive drug and/or alcohol screen

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetic (PK) variables of plasma mycophenolic acid (MPA) and phenolic glucuronide of MPA (MPAG): AUClast, AUCinf, Cmax | Days 1 and 13: predose, and at 0.5, .75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24, 48, 72, and 96 hours postdose
  Area under the concentration-time curve (AUC) from the time of dosing to the last quantifiable concentration (AUClast), AUC from the time of dosing to infinity (AUCinf), and maximum concentration (Cmax)

SECONDARY OUTCOMES:
PK of plasma isavuconazole: Trough concentration (Ctrough) | Day 11, Days 14-16, predose and on Day 17, predose and 24 hours postdose
Composite of PK variables of plasma isavuconazole concentration: AUCtau, Cmax, and tmax | Days 12 and 13: predose and at 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, and 24 hours postdose
  AUC during the time interval between consecutive dosing (AUCtau), time to attain Cmax (tmax)
Composite of PK variables of plasma MPA: tmax, t1/2, Vz/F, and CL/F | Days 1 and 13: predose, and at 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24, 48, 72, and 96 hours postdose
  Apparent terminal elimination half-life (t1/2), apparent volume of distribution (Vz/F), and apparent body clearance after oral dosing (CL/F)
Composite of PK variables of plasma MPAG: tmax and t1/2 | Days 1 and 13: predose, and at 0.5, .75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24, 48, 72, and 96 hours postdose
Safety assessed through the reporting of adverse events, laboratory evaluations, electrocardiograms (ECGs) and vital signs | Through Day 17

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Parexel International, LLC, Glendale, California, United States